CLINICAL TRIAL: NCT03853486
Title: ATHN 9: A Natural History Cohort Study of the Safety, Effectiveness, and Practice of Treatment for People With Severe Von Willebrand Disease (VWD)
Brief Title: ATHN 9: Severe VWD Natural History Study
Status: Active, not recruiting | Type: Observational
Sponsor: American Thrombosis and Hemostasis Network (Network)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: ATHN 9
Record Dates: First submitted 2019-01-11; First posted 2019-02-25 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Von Willebrand Diseases
Keywords: VWF; von Willebrand Disease; VWD; Factor; ATHN 9
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All participants will undergo laboratory evaluation. The remaining specimen volume will be stored and may be used for future research.
  Specimens will be tested as follows:
  * FVIII Activity, VWF Antigen, and the VWF:GPIbM Activity Assay. Reflex testing may include: VWD Type 2B Binding, VWD Type 2N Binding, VWF Propeptide Antigen, and/or VWF Quantitative Multimers
  * Genetic sequence analysis of VWF coding regions and adjacent non-coding regions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ATHN 9 is a natural history study to assess the safety of various Von Willebrand Factor (VWF) regimens for different indications (on-demand, surgery and prophylaxis) in adult and pediatric participants with clinically severe congenital VWD.

DETAILED DESCRIPTION:
The overarching objective of this longitudinal, observational and prospective study is to characterize the safety and effectiveness of factor replacement in participants with clinically severe congenital VWD (VWF:Ag, VWF:GPlbM or VWF:RCo of ≤30% or ≤40% of normal with severe bleeding phenotype defined as requiring recurrent use of factor concentrates) enrolled in the ATHNdataset.

This is a longitudinal, observational cohort study being conducted at up to 30 ATHN-affiliated sites. Participants will be followed for 2 years from time of study enrolment. The total study duration is 3 years.

Safety will be measured by the number of reported events defined by the European Haemophilia Safety Surveillance (EUHASS) program. In addition, although not specifically defined by EUHASS, treatment-emergent side effects of therapy will be included as reportable events including: hypersensitivity/allergic reactions, thrombotic events, VW Factor inhibitor development, treatment-emergent side effects of therapy, transfusion-transmitted infections, malignancy, cardiovascular events, neurological events, unexpected poor efficacy and death.

Secondary objectives of ATHN 9 are:

* to enrich and analyze the data from currently enrolled participants with clinically severe congenital VWD in the ATHNdataset via the collection of laboratory data consisting of a standardized diagnostic battery using an ELISA based VWF activity assay, and genetic sequence analysis of VWF coding regions and adjacent non-coding regions;
* to establish a platform for sub-studies for participants with congenital severe VWD, that are treated with VWF products on demand or have started on or switched to a particular VWF containing product for prophylaxis;
* to evaluate the use of factor replacement as prophylaxis in participants over 6-month time periods;
* to describe bleeding events, changes in overall bleeding and annualized bleeding rate (ABR) over the course of the study as measured by individual bleeding components; and
* to describe real-world effectiveness of VWD treatment as measured by health care utilization and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with severe Von Willebrand Disease with Type 3 VWD or VWF:RCo, VWF:GPlbM or VWF:Ag ≤30% of pooled normal control plasma on more than one occasion;
2. Participants with clinically severe VWD as defined by VWF:RCo, VWF:GPlbM or VWF:Ag ≤40% of normal with severe bleeding phenotype defined as requiring recurrent use of factor concentrates; and
3. Co-enrollment in the ATHNdataset.

Exclusion Criteria:

1. Diagnosis of platelet-type VWD;
2. Diagnosis of acquired VWD (clinical diagnosis based on association with hypothyroidism, lymphoproliferative and myeloproliferative disorders, malignancies and cardiovascular disease, typically aortic stenosis or LVAD).

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: This is a natural history study in which it is anticipated that approximately 130 participants will be enrolled. The study will attempt to enroll a target number of at least 30 participants who are receiving VONVENDI but will not mandate the use of VONVENDI.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2019-06-18 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Reported adverse events from VWF regimens for different indications (on-demand, surgery, and prophylaxis) as measured by EUHASS. | 2 years
  Number of adverse events as measured by EUHASS as well as treatment-emergent side effects of therapy for various Von Willebrand Factor (VWF) regimens for different indications (on-demand, surgery and prophylaxis) in adult and pediatric participants with clinically severe congenital VWD.

SECONDARY OUTCOMES:
Enrich and analyze data collected about AE events as defined by EUHASS using standardized diagnostic battery using an ELISA-based VWF assay. | 3 years
  To enrich and analyze the data from currently enrolled participants with clinically severe congenital VWD in the ATHNdataset via the collection of laboratory data consisting of a standardized diagnostic battery using an ELISA-based VWF assay.
Enrich and analyze data collected about AE events, as defined by EUHASS using genetic sequence analysis of VWF coding regions and adjacent non-coding regions. | 2 years
  To enrich and analyze the data from currently enrolled participants with clinically-severe congenital VWD in the ATHNdataset via the collection of laboratory data using genetic sequence analysis of VWF coding regions and adjacent non-coding regions.
Substudy modules will be developed to evaluate and report on cohorts of study participants who initiate treatment with specific product. | 2 years
  To measure the number of participants taking unique VWF products.
Factor replacement used as prophylaxis. | 3 years
  Report number of particpants using factor replacement as prophylaxis.
Capture bleeding events using the Pictorial Bleeding. Assessment Chart. | 3 years
  The number of participants with bleeding events analyzed over the course of the study.
Capture annualized bleeding rate (ABR) using ISTH BAT Assessment Tool. | 3 years
  The change in the annualized bleeding rate (ABR) for participants over the course of the study by analyzing the number of bleeding events divided by the length of time of the treatment (in years).
Calculate the effectiveness of VWD treatment as measured by health care utilization. | 3 years
  The number of visits/hospitalizations.
Analyze the effectivness of VWD treatment as measured by score on PROMIS questionnaire using the 7 PROMIS domains (depression; anxiety; physical function; pain; fatigue; sleep disturbance; and participation in social roles and activities). | 3 years
  Health-related Quality of Life measured annually by the Patient Reported Outcomes Measurement Information System (PROMIS ®) Profile.
Capture bleeding events using the Pictorial Bleeding Assessment Chart. | 3 years
  The number of participants with bleeding events analyzed over the course of the study.
Capture annualized bleeding rates (ABR) using the Pictorial Bleeding Assessment Chart. | 3 years
  The change in the annualized bleeding rate (ABR) for participants over the course of the study by analyzing the number of bleeding events divided by the length of time of the treatment (in years).
Calculate the success of VWD treatment as measured by health care utilization. | 3 years
  The types of visits/hospitalizations
Capture the effectiveness of VWD treatments using health-related quality of life. | 3 years
  Measure walking ability as part of quality of life using the V-WIQ questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sidonio, MD, Principal Investigator — Emory University / Children's Healthcare of Atlanta; Angela Weyand, MD, Principal Investigator — University of Michigan Hemophilia and Coagulation Disorders
Locations (22):
- United States (22):
  - Center for Inherited Blood Disorders, Orange, California
  - University of Colorado Denver Hemophilia and Thrombosis Center, Aurora, Colorado
  - Connecticut Bleeding and Clotting Disorders Center, Farmington, Connecticut
  - University of Florida Hemophilia Treatment Center, Gainesville, Florida
  - Children's Healthcare of Atlanta/Emory, Atlanta, Georgia
  - Bleeding and Clotting Disorders Institute, Peoria, Illinois
  - Indiana Hemophilia and Thrombosis Center (IHTC), Indianapolis, Indiana
  - Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - University of Michigan Hemophilia and Coagulation Disorders, Ann Arbor, Michigan
  - Children's Hospital of Michigan Hemostasis and Thrombosis Center, Detroit, Michigan
  - Michigan State University Center for Bleeding and Clotting Disorders, East Lansing, Michigan
  - Mayo Comprehensive Hemophilia Center, Rochester, Minnesota
  - Washington University Center for Treatment of Bleeding and Blood Clotting Disorders, St Louis, Missouri
  - Nationwide Children's Hospital Columbus, Columbus, Ohio
  - Oregon Health, Portland, Oregon
  - Pennsylvania Comprehensive Hemophilia and Thrombophilia Program / Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Center of Western Pennsylvania, Pittsburgh, Pennsylvania
  - Rhode Island Hemostasis & Thrombosis Center, Providence, Rhode Island
  - University of Tennessee, University Clinical Health (Memphis), Memphis, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Hemophilia Outreach Center, Green Bay, Wisconsin
  - Versiti - Blood Center of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No